CLINICAL TRIAL: NCT05812183
Title: The Effect of Gastric Sleeve-Induced Weight Loss on Shortness of Breath in Patients with Obesity: a Feasibility Study
Brief Title: Gastric Sleeve-Induced Weight Loss on Shortness of Breath in Obesity
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Conducted an interim analysis on similar data
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); Northwestern University (Other)
Responsible Party: Principal Investigator, Edward Harry Livingston, Professor of Surgery, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-001915
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Dyspnea; Quality of Life
MeSH Terms: conditions — Dyspnea | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Surgery is comapred with medical treatments for obesity. Some of the medical treatments will include treatments using FDA-approved medications
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bariatric surgery (Experimental): Gastric sleeve resection will be performed by experienced surgeons. Postoperative care will follow UCLA's postoperative care pathways for gastric sleeve resection.
  Interventions: Device: Bariatric surgery
- Medical weight loss (Experimental): The medical weight loss intervention will follow the University of California at Los Angeles's (UCLA) Research For Obesity (RFO) standard protocol. Over a period of 12 months, patients in the medical weight loss group will follow a very loc caloric diet (VLCD) at the UCLA RFO program. All study patients will be prescribed a VLCD, an exercise regimen and will participate in group classes on behavioral modification. The caloric intake consists of a commercially prepared meal replacement powder supplying 700-800 cal/day. Each formula packet provides 100kcal and 15g of high biological value protein, and the daily allowance of required minerals and vitamins.
  Interventions: Drug: Medical weight loss

INTERVENTIONS:
Device: Bariatric surgery — Gastric sleeve resection will be performed by experienced surgeons. Postoperative care will follow UCLA's postoperative care pathways for gastric sleeve resection.
  Arms: Bariatric surgery
Drug: Medical weight loss — The medical weight loss intervention will follow UCLA's RFO standard protocol. Over a period of 12 months, patients in the medical weight loss group will follow a very low caloric diet (VLCD) at the UCLA RFO program. All study patients will be prescribed a VLCD, an exercise regimen and will participate in group classes on behavioral modification. The caloric intake consists of a commercially prepared meal replacement powder supplying 700-800 cal/day. Each formula packet provides 100kcal and 15g of high biological value protein, and the daily allowance of required minerals and vitamins. Some patients may recieve adjuvant drug therapy including Orlistat (Xenical, Alli), Phentermine-topiramate (Qsymia), Naltrexone-bupropion (Contrave), Liraglutide (Saxenda), Semaglutide (Wegovy), Tirzepatide (Zepbound) or Setmelanotide (Imcivree).
  Arms: Medical weight loss

SUMMARY:
Most research to date on bariatric surgery outcomes has been about metabolic syndrome, a disorder very effectively treated by bariatric surgery. However, obesity is also associated with many other problems that have received much less attention. Amongst the most troubling of these for patients is dyspnea. Dyspnea results in substantial patient distress that can greatly reduce health-related quality of life. Little is known about the relationship between dyspnea, weight loss, and bariatric surgery. Dyspnea is a complex symptom that may lead to adaptive responses, such as the need to rest as a consequence of even minimal activity or seeking medical attention. The main outcome of the study will be measured using a new state-of-the-science validated HRQOL measure, the Patient Reported Outcome Measuring Information System for Heart Failure (PROMIS+HF 27).

DETAILED DESCRIPTION:
The main purpose of this prospective matched cohort study is to determine the feasibility for a future, novel large-scale study, clinical trial that will aim to determine how common dyspnea is in obese patients, how much dyspnea affects their quality-of-life, and how these parameters are affected by medically or surgically induced weight loss. Our basic assumption is that dyspnea is more common than is commonly believed in obese patients and that it profoundly affects quality of life. Our main hypothesis is that weight loss improves dyspnea and HRQOL and that bariatric surgery induced weight loss is more effective than medical weight loss at improving dyspnea-related quality-of-life.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age.
2. All patients undergoing gastric sleeve resection for serious obesity at the Ronald Reagan medical center will be considered for enrollment in the experimental group.
3. English/Spanish speakers.
4. The patients included will be with preserved cognition and a capacity to understand questionnaires.
5. Written informed consent (and assent when applicable) obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Serious cardiovascular disease, previous gastrointestinal surgery, psychological concerns (mental disorders and dementia), recently hospitalized, pulmonary diseases, renal failure, or history of malignancy.
2. Undergoing procedures other than gastric sleeve resection or are having these operations after they have had other bariatric procedures.
3. Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or the quality of the data.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-09 (Actual); Primary Completion 2025-02-12 (Estimated); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Dyspnea | 12 months
  Will be assessed using the PROMIS+HF 27 will be administered via RedCap for patients both groups.
  PROMIS+HF 27 is part of a National Institutes of Health initiative to develop state-of-the art measures for quality of life. PROMIS+HF 27 contains 3 questions about dyspnea severity. Each of them can be assessed individually or the 3 combined to increase measurement precision into a dyspnea severity domain score.

SECONDARY OUTCOMES:
Health related quality of life | 12 months
  Will be assessed using the PROMIS+HF 27 will be administered via RedCap for patients both groups.
  PROMIS+HF 27 is part of a National Institutes of Health initiative to develop state-of-the art measures for quality of life.

IPD SHARING:
Plan to Share IPD: No